CLINICAL TRIAL: NCT00745706
Title: Discerning Symptomatic and Asymptomatic Episodes Pre and Post Radiofrequency Ablation of Atrial Fibrillation
Acronym: DISCERN-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, David Birnie, M.D., Director of Arrythmia Service, Ottawa Heart Institute Research Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UOHI-01
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Other): Implantable Loop Recorder (ILR) implant
  Interventions: Device: Implantable Loop Recorder (ILR)

INTERVENTIONS:
Device: Implantable Loop Recorder (ILR) — Insertion of ILR 3 months prior to clinical ablation procedure to collect data on actual Atrial Fibrillation episodes and correlation with patient symptoms through patient diary entry. Then patient undergoes their previously indicated clinical ablation procedure and is then followed up with ILR insitu for 30 months post-ablation for the same as mentioned above.
  Other Names: Reveal XT

SUMMARY:
Atrial Fibrillation (AF) is a common heart rhythm problem that can be eliminated by a radiofrequency ablation procedure. The purpose of this study is to assess the amount of AF that occurs before and after an ablation procedure associated with symptoms versus AF that is not associated with any symptoms. This study will confirm whether patients' symptoms or lack of symptoms post-ablation correlate well with actual episodes of Atrial Fibrillation. This is important information for physicians to know as it will help guide patient care post-ablation in the future. Information on patients' AF episodes will be collected by an implantable loop recorder (ILR) which will be implanted in all study patients 3 months prior to their AF ablation procedure. The ILR will automatically collect information on detected AF episodes while patients will records any symptoms related to AF episodes in study diaries.

DETAILED DESCRIPTION:
Patients scheduled to undergo a first time ablation for AF will be implanted with an implantable loop recorder (ILR), capable of automatically recording episodes of AF, 3 months prior to their ablation procedure. Patients will also be given a standardized diary in which they will record all perceived episodes of AF. Patients will have the data from the ILR downloaded prior to their ablation to record baseline AF data.

A blanking period of 3 months will be used to censor early recurrences post-ablation. A 'successful' AF ablation will be defined as a lack of AF episodes > 2min at least 3 months post-ablation. A 'Failure' AF ablation will encompass all patients not meeting the definition of 'success'. Redo ablation procedures will be allowed in this protocol for patients who continue to have AF recurrences beyond the first three months post-ablation.

After the patient's ablation procedure, patients will be followed every 3 months for 18 months. At each follow-up visit data on AF episodes from the ILR and the patient diaries will be collected. Patients will be blinded to the data downloaded from the device.

Further data will be collected as the patient study follow-up period has been extended to include a 30-month post-ablation visit with device interrogation as device battery is 36-42 months.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old.
* First-time ablation procedure for AF.
* Symptomatic AF which has been refractory to at least one antiarrhythmic medication. "Symptomatic" patients should be patients who feel that they are aware of when they are in or out of AF. Symptoms may include palpitations, shortness of breath, chest pain, fatigue, or other symptoms, or any combination of the symptoms listed above.
* Patients must have paroxysmal or persistent AF. Paroxysmal patients should have had at least 4 episodes of AF in the 6 months prior to assessment/ablation. Paroxysmal AF is defined as AF which spontaneously terminates within 7 days. Persistent AF is defined as AF which sustains for longer than 7 days, or AF lasting less than 7 days which requires either pharmacologic or electrical cardioversion.
* At least one episode of AF must have been documented by ECG or Holter within 12 months of inclusion in the study.
* No contraindication to systemic anticoagulation with heparin or coumadin.
* Patients must be able and willing to provide written informed consent to participate in the study.

Exclusion Criteria:

* Patients with permanent atrial fibrillation. Permanent AF is defined as chronic, persisting AF (typically more than 1 year) for which cardioversion (pharmacologic or electrical) has failed or will never be attempted.
* Patients with AF felt to be secondary to an obvious reversible cause.
* Patients with contraindications to systemic anticoagulation with heparin or coumadin.
* Patients who have previously undergone atrial fibrillation ablation.
* Patients who are or may potentially be pregnant.
* Left atrial size > or equal to 55 mm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-09; Primary Completion 2014-04 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Incidence of asymptomatic versus symptomatic AF pre-ablation | 3 months
Incidence of asymptomatic versus symptomatic AF recurrence > 3months post-AF ablation in patients with "success" after ablation. | 30 months
Incidence of asymptomatic versus symptomatic AF recurrence > 3 months post-AF ablation in patients with "failure" after ablation | 30 months

SECONDARY OUTCOMES:
Incidence of peri-procedural and post-procedural embolic events | 24 hours
Correlation of early recurrences (<3 months post-ablation) to late recurrences (> 3 months post-ablation) | 3-30 months
Incidence of very late AF recurrence (beyond 12 months psot-ablation) in "successful" patients post-ablation (determined both by AF episodes and burden) | 30 months
Comparison of "success" and "failure" rates as determined by ILR versus traditional, clinically-indicated ECG and holter monitoring | 30 months
Cost-effectiveness analysis of using ILR monitoring for post-AF ablation monitoring versus traditional follow-up (ECGs, holter, loop recorders) | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Atul Verma, M.D., Principal Investigator — Southlake Regional Health Centre; David Birnie, M.D., Principal Investigator — Ottawa Heart Institute Research Corporation; Paul Novak, M.D., Principal Investigator — Royal Jubilee Hospital
Locations (8):
- Canada (8):
  - Victoria Cardiac Arrhythmia Trials Inc., Victoria, British Columbia
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Hôpital Général de Montréal-McGill, Montreal, Quebec
  - Hôpital Laval, Québec, Quebec

REFERENCES:
- [Result] Verma A, Champagne J, Sapp J, Essebag V, Novak P, Skanes A, Morillo CA, Khaykin Y, Birnie D. Discerning the incidence of symptomatic and asymptomatic episodes of atrial fibrillation before and after catheter ablation (DISCERN AF): a prospective, multicenter study. JAMA Intern Med. 2013 Jan 28;173(2):149-56. doi: 10.1001/jamainternmed.2013.1561. PMID 23266597